CLINICAL TRIAL: NCT06095869
Title: Ege University Faculty of Health Sciences Midwifery Department
Brief Title: Progressive Relaxation Exercises,Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, çigdem gök, specialist midwife, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: EGE-C-GOK-001
Record Dates: First submitted 2023-06-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Progressive Relaxation Exercises
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- progressive relaxation exercise group (Experimental): intervention group with progressive relaxation exercise
  Interventions: Other: progressive relaxation exercise; Other: relaxation background music; Other: control group
- relaxation background music group (Experimental): intervention group with relaxation background music
  Interventions: Other: progressive relaxation exercise; Other: relaxation background music; Other: control group
- control group (Experimental): group receiving routine health protocol and no intervention
  Interventions: Other: progressive relaxation exercise; Other: relaxation background music; Other: control group

INTERVENTIONS:
Other: progressive relaxation exercise — Breastfeeding mothers in the progressive relaxation exercise group were applied gradual relaxation exercise before going to bed 3 days a week and for 4 weeks, under the supervision of the researcher, accompanied by a training CD prepared by the Turkish Psychologists Association.
Other: relaxation background music — In the relaxation background music group, breastfeeding mothers were listened to relaxation background music on the Progressive Relaxation Exercise CD before going to bed 3 days a week and for 4 weeks.
Other: control group — Mothers in this group received routine care practices in the clinic. No intervention was made to the mothers in the control group, only data collection tools were applied.

SUMMARY:
OBJECTIVE: The research was conducted to examine the effects of progressive relaxation exercises on mothers' breastfeeding status, self-efficacy and maternal attachment level.

DETAILED DESCRIPTION:
may 2022 and November 2022. The sample of the study consisted of 114 mothers who were breastfeeding in the postpartum period. In the study, 38 breastfeeding mothers were included in the PGE, GFM and control groups. Breastfeeding mothers in the PGE group were given a PGE application 3 days a week before going to bed and for 4 weeks, accompanied by a training CD prepared by the Turkish Psychological Association, under the supervision of the researcher. On the other hand, the breastfeeding mothers in the GFM group were listened to the relaxation background music included in the Progressive Relaxation Exercise CD 3 days a week before going to bed and for 4 weeks. Mothers in the control group received routine care practices applied in the clinic. The mothers in the control group did not receive any intervention and only measurement tools were applied. 'Personal Information Form', 'Breastfeeding Self-Efficacy Scale' and 'Maternal Attachment Scale', 'Visual Analog Scale', 'Breastfeeding Classification' were used to collect data. Standard Deviation, Mean, Frequency and Chi-square tests were used to evaluate the data. Analysis of variance was used for repetitive measurements for the evaluation of breastfeeding self-efficacy and maternal attachment level within the group, and one-way analysis of variance was used for the evaluation between groups.

ELIGIBILITY:
Inclusion Criteria:Mothers over the age of 18,

* At least primary school graduate, able to read and understand Turkish,
* Has a phone and internet
* Has an only and healthy baby,
* Does not have a condition that prevents him from doing PGE,
* The baby was born between 2500-4000 g,
* Those who live within the provincial borders of Uşak,
* No hearing problem,
* Mothers of babies who do not have sucking problems (cleft palate-lip, frenilium, galactosemia, prematurity),
* Mothers who do not have any health problems affecting breastfeeding (mastitis, breast abscess, nipple crack, candida albicans, flat and sunken nipples, Wilson's disease in the mother, an active disease of the mother that prevents breastfeeding, and drug use),
* Mothers without musculoskeletal disorders, The mothers who volunteered to participate in the study.

Exclusion Criteria:

* Practicing relaxation exercises before
* Mothers using chronic opioids, antidepressants and psychoactive drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-04 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in breastfeeding self-efficacy score averages change in breastfeeding self-efficacy scores | in the first two weeks postpartum, in the 1st and 2nd months after birth
  To determine the breastfeeding self-efficacy score averages, the breastfeeding self-efficacy scale average scores were compared, and the breastfeeding self-efficacy scale was applied to the mothers.The scale assessing breastfeeding self-efficacy is a 5-point Likert type (1 = Not at all sure, 2 = Very unsure, 3 = Sometimes sure, 4 = Sure, 5 = Very sure). All items of the scale have a positive meaning. The highest score that can be obtained from the scale is 70 and the lowest score is 14. The scale has no cut-off point. Increasing scores on the scale indicate high breastfeeding self-efficacy.

SECONDARY OUTCOMES:
change in maternal attachment score averages | postpartum 1st month and 2nd months after birth
  To determine the maternal attachment mean scores, the maternal attachment mean scores were compared and the maternal attachment scale was applied to the mothers.Each item ranges from "always" to "never" and is a 4-point Likert-type scale. It is calculated as always (a) = 4 points, often (b) = 3 points, sometimes (c) = 2 points and never (d) = 1 point, and each item contains direct expressions. The lowest score obtained from the scale varies between 26 and the highest score 104. The higher the score obtained from the scale, the higher the maternal attachment is considered to be.

OTHER OUTCOMES:
change in breastfeeding status | in the first two weeks postpartum, in the 1st and 2nd months after birth
  To evaluate the breastfeeding status of mothers, a form evaluating the breastfeeding status prepared by the World Health Organization in 1991 was used.
satisfaction rating | postpartum 4th month
  A satisfaction scale was applied to evaluate the satisfaction of mothers with the interventions applied.This form, prepared by the researcher within the scope of the literature; It consists of five questions that evaluate how effective the application is for mothers in the PGE and GFM groups, how satisfied they are with the application, and whether they would recommend it to other mothers.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Health Sciences Midwifery Department, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No